CLINICAL TRIAL: NCT03540745
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Nexalin Electrical Brain Stimulation as an Adjunctive Therapy for Substance Dependence
Brief Title: Nexalin Therapy as a Viable Adjunctive Treatment for Substance Use Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Carrier Clinic (Other)
Responsible Party: Principal Investigator, Michael A. Grandner, Assistant Professor of Psychiatry, Psychology, and Medicine Director, Sleep & Health Research Program, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1712118546
Record Dates: First submitted 2018-03-12; First posted 2018-05-30 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Depression; Anxiety; Insomnia; Substance Abuse
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with block randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and investigators are blind to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TES Treatment (Experimental): Where subject is randomized to TES.
  Interventions: Device: TES Treatment
- TES-SHAM Treatment (Placebo Comparator): Where subject is randomized to a SHAM condition
  Interventions: Device: TES-SHAM Treatment

INTERVENTIONS:
Device: TES Treatment — Device: Nexalin Based Trans-Cranial Electrical Stimulation The Nexalin device, FDA clearance (501K=K024377, Classification: Stimulator, Cranial Electrotherapy: CFR 882. 5800: U.S. Patent #6904322B2), produces a square waveform that provides trans-cranial electrical stimulation to the brain delivered at a frequency of 77.5 Hz at 0 to 4 mA peak current. Other Name: TES
  Arms: TES Treatment
Device: TES-SHAM Treatment — Device: Nexalin Based Trans-Cranial Electrical Stimulation The Nexalin device, FDA clearance (501K=K024377, Classification: Stimulator, Cranial Electrotherapy: CFR 882. 5800: U.S. Patent #6904322B2), produces a square waveform that provides trans-cranial electrical stimulation to the brain delivered at a frequency of 77.5 Hz at 0 to 4 mA peak current. Other Name: TES
  Arms: TES-SHAM Treatment

SUMMARY:
The purpose of this research study is to determine whether Nexalin Trans-cranial Electrical Stimulation (TES) is a viable adjunctive treatment of substance use treatments.

DETAILED DESCRIPTION:
A Randomized Controlled Trial with block randomization. Inpatient subjects actively seeking substance abuse treatment at the Carrier Clinic who are diagnosed with a substance use disorder, including alcohol use disorder, tobacco use disorder, polysubstance use disorder, or other substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide informed consent, assessed by the study clinician
2. Be able to speak, read and write fluently in English, assessed by the study clinician
3. Be committed to completion of the study. The subject will need to attest to availability for 10 to 15 treatments over a 5 to 8 day period for the treatment protocol.
4. Be adults over age 18 and under age 65
5. Be actively receiving substance use treatment for a substance use disorder

Exclusion Criteria:

1. Pregnant or at risk of becoming pregnant
2. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, might confound the interpretation of the study results, or put the person at undue risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 5-8 Days
  Reduction in depressive symptoms as a result of Nexalin vs Sham

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Grandner, PhD, Principal Investigator — University of Arizona
Locations (1):
- Carrier Clinic, Belle Mead, New Jersey, United States